CLINICAL TRIAL: NCT03010202
Title: Prolonging the Response by Low-dose Rituximab Maintenance Therapy in Immune Thrombocytopenia: a Randomized Placebo-controlled Trial - the PROLONG Trial
Brief Title: The PROLONG Trial - Rituximab Maintenance Therapy in ITP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); University Hospital of North Norway (Other); Haukeland University Hospital (Other); Odense University Hospital (Other); Centre Hôpital Universitaire Farhat Hached (Other); Henri Mondor University Hospital (Other); University Hospital, Akershus (Other); Cairo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGCH004
Record Dates: First submitted 2016-12-28; First posted 2017-01-04 (Estimated); Last update posted 2024-05-29 (Actual); Status verified 2023-11

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic
Keywords: immune thrombocytopenia; rituximab; thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — Dexamethasone; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Induction phase: Rituximab+Dexamethasone (Experimental): Open-label, intravenous infusions of rituximab 1000 mg and oral dexamethasone 20 mg daily for 4 days given on day 1 and day 15.
  Interventions: Drug: Dexamethasone
- Induction phase: Rituximab (No Intervention): Open-label, intravenous infusions of rituximab 1000 mg given on day 1 and day 15.
- Maintenance phase: Rituximab (Experimental): Patients who respond to rituximab in the induction phase will be proceed into the maintenance phase and randomized to rituximab infusion of 500 mg in week 1 and week 24, or
  Interventions: Drug: Rituximab
- Maintenance phase: Placebo (No Intervention): Infusion of normal saline 0,9% in week 1 ande week 24 in second randomization.

INTERVENTIONS:
Drug: Dexamethasone — Comparing the effect of Rituximab infusion With or without Dexamethasone
  Arms: Induction phase: Rituximab+Dexamethasone
Drug: Rituximab — Comparing maintenance dose of 500mg Rituximab at week 1 and week 24 to Placebo
  Other Names: Mabthera
  Arms: Maintenance phase: Rituximab

SUMMARY:
This study is a two phase study that aims to evaluate if low-dose Rituximab maintenance therapy may prolong the the effect of Rituximab in immune thrombocytopenia.

DETAILED DESCRIPTION:
This is a multi-center, international, randomized, two-phase study:

First phase (induction phase) is open-label, hypothesis-generating, involving 1:1 randomization into: rituximab (group 1) or rituximab plus dexamethasone (group 2) to determine if the response to rituximab can be improved by the addition of dexamethasone.

Second Phase (maintenance phase) is the main part of the study, involving 1:1 double-blind randomization into low dose rituximab or placebo to determine if the response achieved in the first phase can be prolonged by administrating maintenance treatment with low dose rituximab.

Primary objective:

To determine if maintenance therapy with low-dose rituximab is superior to placebo in prolonging responses among ITP patients who achieved an initial response with rituximab.

Secondary objectives:

1. To explore if the initial overall response rate, at week 24, can be improved by at least 10% by adding dexamethasone to rituximab (induction phase).
2. To assess the safety of study treatment, especially infectious episodes (induction & maintenance phases).
3. To assess bleeding complications during the study (induction & maintenance phases).
4. To assess the use of rescue medications and other platelet-elevating therapies during the study (induction & maintenance phases).
5. To determine rate of Complete Response (CR) during induction phase and sustained CR during maintenance phase (induction & maintenance phases).
6. To determine the duration of overall response and CR (induction & maintenance phases).
7. To assess health-related quality of life and fatigue (induction & maintenance phases).

ELIGIBILITY:
Inclusion Criteria First randomization (Induction phase):

1. Male or female aged ≥18 years.
2. Diagnosis of primary ITP of less than one year duration having a platelet count of ≤ 30 x109/L measured within 4 weeks prior to inclusion with failure to achieve initial response or relapse either after one cycle of dexamethasone (40 mg daily for 4 days) or 4 weeks with any other steroid (prednisone or prednisolone). Platelet count between 31 to 50 x109/L is accepted if higher platelet count is required due to concomitant antiplatelet therapy or bleeding.
3. Scheduled intravenous treatment of rituximab.
4. Signed and dated written informed consent.
5. Females of child-bearing potential accepting to follow effective contraceptive methods for at least 12 months following the last administration of rituximab or placebo.

Inclusion criteria second randomization (maintenance phase):

1. Completion of the induction phase (phase 1) of the study.
2. Sustained response at the end of phase 1.
3. Randomization within 4 weeks after the completion of phase 1, i.e. between week 24 and 28.

Exclusion Criteria first randomization (Induction phase):

1. Previous treatment for ITP with: rituximab, other immune suppressants (including mycophenolate mofetil, aziothioprin, cyclosporine), chemotherapy or splenectomy.
2. Pregnancy or lactation.
3. Known active gastro-duodenal ulcer.
4. Secondary ITP: ITP associated with lymphoma, chronic lymphocytic leukemia, autoimmune disorders such as, common variable immune deficiency, human immunodeficiency virus, or hepatitis C or thrombocytopenia associated with myeloid dysplasia.
5. Concomitant autoimmune hemolytic anemia.
6. History of any major cardiovascular event within the 6 months prior to randomization, including but not limited to: myocardial infarction, unstable angina, cerebrovascular accident, or New York Heart Association Class III or IV heart failure.
7. Active hepatitis B virus or patients with positive HBsAG or HBcAB.
8. Patients with active severe infection, including systemic mycotic infections or a history of recurring or chronic infections or with underlying conditions which may further predispose patients to serious infection.
9. Known allergy and/or sensitivity or contraindication to rituximab or dexamethasone or any of the ingredients.
10. Patients in a severely immune compromised state.
11. Known contraindication to a treatment with any proton-pump inhibitor.
12. Active malignancy or history of malignant disease during the last 2 years except cured skin cancer.
13. Patients with history of poor compliance or history of alcohol/drug abuse or excessive alcohol beverage consumption that would interfere with the ability to comply with the study protocol, or current or past psychiatric disease that might interfere with the ability to comply with the study protocol or give informed consent.

Exclusion criteria second randomization (maintenance phase) 14. Severe allergic reaction or serum sickness due to rituximab in phase 1 of the study.

15. Pregnancy. 16. Treatment with rescue medication after week 18. 17. Patients refusing to continue in the study (withdrawal of consent). 18. Splenectomy performed for any cause.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2016-12; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Sustained of overall response | 52 weeks
  sustained overall response during maintenance phase [loss of overall response is defined as: (1) two consecutive measurements with platelet counts < 50 x 109/L taken at 1-8-week interval, and/or, (2) use of any ITP-directed therapies, other than study medication, because of bleeding or thrombocytopenia, except for preoperative elevation of platelet count] (this endpoint applies to maintenance phase only).

SECONDARY OUTCOMES:
Improvement at overall response rate in week 24 | Week 24 (+/- 2 weeks)
  Overall response during induction phase defined as mean platelet count, determined in week 24 (± 2 weeks) after induction therapy, > 50 x 10E9/L , without use of any other ITP-directed therapies after week 12 following the first randomization (this endpoint applies to induction phase only).
Safety assessed by the frequency of > grade II adverse events (this endpoint applies to both phases) | 24 weeks and 52 weeks
  Safety assessed by the frequency of > grade II adverse events (this endpoint applies to both phases).
Grade of bleeding during the study (during both phases) | 24 weeks and 52 weeks
  Grade of bleeding (this endpoint applies to both phases).
Sustained Complete Response (CR) during maintenance phase | 52 weeks
  Sustained Complete Response (CR) during maintenance phase defined as platelet count > 100 x 109/L maintained during maintenance phase, without the use of any ITP-directed therapies
Complete Response during induction phase | 24 weeks (+/- 2 weeks)
  Complete Response (CR) during induction phase defined as platelet count, determined in week 24 (± 2 weeks), > 100 x 109/L without use of any other ITP-directed therapies after week 12 following the first randomization (induction phase)
Rescue medication or other elevating platelet therapy | after 12 weeks in induction phase and 40 weeks in maintenance phase
  Administration of rescue medication or other elevating platelet therapy
  1. After week 12 (induction phase)
  2. During maintenance phase (maintenance phase).
Platelet count Levels > 50 x 109/L during maintenance phase | phase 2 (52 weeks)
  Percentage of patients with more than 80% of platelet counts level > 50 x 109/L during the maintenance phase (this endpoint applies to maintenance phase only).
Health related quality of life | First phase at 24 weeks and second phase at 52 weeks
  Health-related quality of life assessed by SF-36 questionnaire (this endpoint applies to both phases).

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Ghanima, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (1):
- Ostfold Hospital Trust, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: No